CLINICAL TRIAL: NCT06122311
Title: Drug Nephrotoxicity Amelioration in Hematological Malignancies Patients by N-acetylcysteine
Brief Title: Drug Nephrotoxicity Amelioration by N-acetylcysteine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Yasmin medhat munir Mohamed, Teaching assistant, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANP
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Drug-Induced Nephropathy
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Intervention and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): amphotericin b (0.5-1.25 mg/kg )over 6-8 hours +NAC 600mg twice daily throughout amphotericin b treatment
  Interventions: Drug: N Acetylcysteine
- amphotericin b (No Intervention): amphotericin b (0.5-1.25mg/kg)over 6-8 hours infusion

INTERVENTIONS:
Drug: N Acetylcysteine — N-acetylcysteine sachets 600 mg twice daily
  Other Names: Acetylcysteine
  Arms: N-acetylcysteine

SUMMARY:
When treating individuals with febrile neutropenia, amphotericin B (AmB-d) is one of the most effective treatments against often fatal systemic fungal infections.Nephrotoxicity from amphotericin B can develop with an incidence of up to 80.This emphasizes the value of nephroprotectant agent use.Because of N-acetylcysteine's antioxidant, antiapoptotic, vasodilator properties and its therapeutic effects on contrast nephropathy. Acetylcysteine's impact on amphotericin B-induced nephrotoxicity in cancer patients is assessed.

DETAILED DESCRIPTION:
Severe fungal infections continue to be a significant source of morbidity and mortality in haematology units despite recent therapeutic advancements. The first anti-fungal medication that was successful against systemic mycoses was characterised as the traditional amphotericin B in the middle of the 1950s.AMB remains the treatment of choice for many serious fungal infections in vulnerable hosts owing to its excellent spectrum of activity and its low resistance rates. To date, it continues to be the agent with the widest spectrum of action and the lowest resistance potential of any known antifungal agent.In spite of clinical effectiveness, AmB treatment is associated with a range of acute and chronic adverse reactions . Nephrotoxicity and consequent electrolytes imbalances have been demonstrated as the most clinically significant adverse reaction of AmB that can restrict its clinical utility. Up to 80 % of AmB recipients during the first two weeks of treatment may develop some degree of reversible kidney injury . In addition, nearly 15 % of these patients may require dialysis which can lead to prolongation of hospital stay, increased total treatment costs, and mortality .

N-acetylcysteine, a drug with vasodilating, antiapoptotic, and anti-oxidant features, has been found to diminish the nephrotoxicity of cisplatin , cyclosporine and gentamicin . The results of two experimental studies in rats have suggested that N-acetylcysteine can mitigate GFR reduction as well as renal tubular apoptosis caused by AmB .

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years.
* Patients who have indication for systemic (injection) for conventional amphotericin at least 7 days.

Exclusion Criteria:

* documented acute kidney injury defined by an increase in serum creatinine ‡ 0.3 mg/dl within 48 h, or an increase in serum creatinine by ‡ 1.5 times baseline within the prior 7 days, or urine volume <0.5 ml/kg/h for 6 h
* documented chronic kidney disease (clearance creatinine below 60 ml/min/1.73 m2 calculated by the abbreviated Modification of Diet in Renal Disease equation), history of peritoneal or hemodialysis for > 3 months
* sepsis
* Severe hemorrhage(Blood loss > 3 litres)
* Patient with cardiac or chronic liver disease history of receiving AmB by any administration route within the recent 14 days known allergy to either amphotericin b or N-acetylcysteine.
* receiving any formulation of NAC within the last week.
* unable to tolerate oral intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
incidence of nephrotoxicity | During the intervention
  minimum of 0.3 mg/dL increase in serum creatinine within 48 hours from amphotericin B initiation.

SECONDARY OUTCOMES:
electrolyte imbalances | During the intervention
  Hypokalemia and hypomagnesemia were defined as serum potassium levels less than 3 mEq/L and serum magnesium levels less than 1.2 mEq /L, respectively.

OTHER OUTCOMES:
cost effectiveness analysis | From start of amphotericin b to discharge or death ,whichever came first or up to 120 days
  incremental cost effectiveness ratio
length of hospital stay(days) | From start of amphotericin b to discharge or death ,whichever came first or up to 120 days
  duration a patient spends in a hospital

CONTACTS AND LOCATIONS:
Overall Officials: yasmin munir, master, Principal Investigator — Helwan University
Locations (1):
- Helwan University, Cairo, Egypt

REFERENCES:
- [Background] Karimzadeh I, Khalili H, Sagheb MM, Farsaei S. A double-blinded, placebo-controlled, multicenter clinical trial of N-acetylcysteine for preventing amphotericin B-induced nephrotoxicity. Expert Opin Drug Metab Toxicol. 2015;11(9):1345-55. doi: 10.1517/17425255.2015.1042363. Epub 2015 Jun 11. PMID 26050706
- [Background] Odabasi Z, Karaalp A, Cermik H, Mohr J, Tigen ET, Koc M, Korten V. Reduction of amphotericin B-induced renal tubular apoptosis by N-acetylcysteine. Antimicrob Agents Chemother. 2009 Jul;53(7):3100-2. doi: 10.1128/AAC.00001-09. Epub 2009 May 4. PMID 19414577
- [Background] Feldman L, Efrati S, Dishy V, Katchko L, Berman S, Averbukh M, Aladjem M, Averbukh Z, Weissgarten J. N-acetylcysteine ameliorates amphotericin-induced nephropathy in rats. Nephron Physiol. 2005;99(1):p23-7. doi: 10.1159/000081799. PMID 15637469
- [Derived] Ebid AIM, Mohamed HS, Mohammed YMM, Mohamed Abdel Motaleb SM. Efficacy, Safety, and Cost-Effectiveness of N-Acetylcysteine in Preventing Amphotericin B Nephrotoxicity in Egyptian Patients with Hematological Malignancies: A Randomized Controlled Trial. Hosp Pharm. 2025 May 6:00185787251337615. doi: 10.1177/00185787251337615. Online ahead of print. PMID 40342610